CLINICAL TRIAL: NCT03389503
Title: Comparison Between Left and Right Transradial Approach During Coronary Angiography and Percutaneous Coronary Intervention
Brief Title: Comparison of Left and Right Transradial Approach for CAG and PCI
Acronym: COMPARE-Rad
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Young Jin Youn, Assistant professor, Wonju Severance Christian Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CR316096
Record Dates: First submitted 2017-12-27; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Coronary Artery Disease; Stable Angina; Unstable Angina; Non-ST Elevation Myocardial Infarction; ST-segment Elevation Myocardial Infarction; Ischemic Heart Disease Without Angina
Keywords: Access site; Transradial access; Coronary artery disease; Learning curve
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable; Angina, Unstable; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: 1~3 months: Right radial approach 4~6 months: Left radial approach
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right radial approach (Active Comparator): Right radial approach for coronary angiography and coronary intervention
  Interventions: Procedure: Radial approach
- Left radial approach (Active Comparator): Left radial approach for coronary angiography and coronary intervention
  Interventions: Procedure: Radial approach

INTERVENTIONS:
Procedure: Radial approach — Approach site for coronary angiography and coronary intervention

SUMMARY:
This trial will compare the procedural success rate between right and left radial approach in patients undergoing coronary angiography and coronary intervention.

DETAILED DESCRIPTION:
The three operators who are proficient in the left radial approach for coronary angiography and coronary intervention will be assigned to the right radial approach for 3 months (phase 1). After then, these three operators will switch approach site to the left radial for another 3 months (phase 2).

Procedural success, time of the procedure, use of contrast agent, and fluoroscopic data will be compared between right radial approach (phase 1) group and left radial approach (phase 2).

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing coronary angiography via radial approach
* Subjects undergoing coronary intervention via radial approach
* Subjects give written informed consent

Exclusion Criteria:

* Subjects undergoing procedure(s) other than coronary angiography or intervention
* Subjects with contraindication of radial approach (i.e, non-palpable radial pulsation, abnormal Allen's test, known radial artery tortuosity or occlusion, arteriovenous fistula for dialysis)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2017-09-07 (Actual)

PRIMARY OUTCOMES:
Procedural success | At the end of procedure
  Finishing coronary angiography/intervention without changing approach site

SECONDARY OUTCOMES:
Puncture time | At the end of procedure
  Duration from the start of local anesthesia infiltration to the insertion of sheath
Coronary angiography time | At the end of procedure
  Duration from the insertion of sheath to the end of coronary angiography
Puncture + Coronary angiography time | At the end of procedure
  Sum of puncture time and coronary angiography time
Coronary intervention time | At the end of procedure
  Duration from the end of coronary angiography to the end of coronary intervention
Contrast amount during coronary angiography | At the end of procedure
  Amount of contrast agent used during coronary angiography
Contrast amount during coronary intervention | At the end of procedure
  Amount of contrast agent used during coronary intervention
Fluoroscopic dose, dose area product during coronary angiography | At the end of procedure
  Dose area product during coronary angiography
Fluoroscopic dose, dose area product during coronary intervention | At the end of procedure
  Dose area product during coronary intervention
Fluoroscopic time during coronary angiography | At the end of procedure
  Fluoroscopic time during coronary angiography
Fluoroscopic time during coronary intervention | At the end of procedure
  Fluoroscopic time during coronary intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No